CLINICAL TRIAL: NCT01860664
Title: Phase 2 EFFICACY AND SAFETY OF HYDROCORTISONE OPHTHALMIC OINTMENT - VERSUS PLACEBO IN THE TREATMENT OF ALLERGIC CONJUNCTIVITIS
Brief Title: Hydrocortisone Ophthalmic Ointment 0.5% for Treatment of Allergic Conjunctivitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The Sponsor has stopped responding to calls and emails
Sponsor: Koffler Vision Group (Other)
Collaborators: Fera Pharmaceuticals, LLC (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F2012-05
Record Dates: First submitted 2013-05-20; First posted 2013-05-23 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Allergic Conjunctivitis
Keywords: allergy; allergic; conjunctivitis; corticosteroid; hydrocortisone; ophthalmic; ointment
MeSH Terms: conditions — Conjunctivitis, Allergic; Hypersensitivity; Conjunctivitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- hydrocortisone ophthalmic ointment 0.5% (Experimental): Topical ophthalmic corticosteroid ointment, is produced in a concentration of 0.5% of hydrocortisone Acetate in a vehicle composed of mineral oil and white petrolatum
  Interventions: Drug: hydrocortisone ophthalmic ointment 0.5%
- Placebo (Placebo Comparator): mineral oil and white petrolatum
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: hydrocortisone ophthalmic ointment 0.5% — * Patients will be instructed to apply Hydrocortisone Ophthalmic Ointment 0.5% or placebo in the lower cul de sac or lid margin BID
  * Patients will be instructed to not use the study medications at least 2 hours prior to their appointment.
  * Study medication dosing details:
    * 0.05 grams hydrocortisone per gram of combination product
    * each application equal to 1/20th of a gram
    * total amount of active ingredient applied to each eye per application = 0.0025 grams hydrocortisone
    * total amount hydrocortisone applied per eye per day = 0.005 grams hydrocortisone
    * Total amount of active ingredient applied per eye throughout duration of the two week study = 0.07 grams hydrocortisone
  Other Names: PF01335
  Arms: hydrocortisone ophthalmic ointment 0.5%
Drug: placebo — Mineral oil and white petrolatum
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of hydrocortisone ophthalmic ointment compared to placebo in the treatment of Allergic Conjunctivitis.

DETAILED DESCRIPTION:
Compare the safety and efficacy of Hydrocortisone Ophthalmic Ointment 0.5% vs. Placebo for the reduction of signs and symptoms associated with allergic conjunctivitis. Demonstration of efficacy is a statistically significant improvement in itching on a 0 to 4 patient subjective assessment itch score compared to the vehicle arm and at least a 25% (or 1 full unit or more) improvement in itch scores. Efficacy for bulbar redness scores would be indicated by a statistically significant improvement in redness on a zero to 4 based on the investigators objective assessment compared to the vehicle group. Differences of at least 25% on the four point scale would be considered clinically significant when attained at the majority of time points.

ELIGIBILITY:
Inclusion Criteria

a) Diagnosis of allergic conjunctivitis. b) Must be at least 18 years of age c) Must be able and willing to comply with all treatment and follow up procedures d) Best corrected visual acuity of 0.3 logMAR or better (Snellen equivalent score of 20/40 or better) in each eye at Visit 1 e) Conjunctival redness score ≥1.5 in at least one eye at Visit 1 f) Subject reported itching assessment >2.0 in at least 1 eye at Visit 1 g) Mean IOP >8 and <24 in each eye h) If female of childbearing potential, are non-lactating and non-pregnant, and must be willing to use an approved birth control method for the duration of the study, and must have a negative urine pregnancy test. (Urine pregnancy test will be conducted at Visit 1 after subject completes Informed Consent Document prior to any study procedures being performed.) 5.4 Exclusion Criteria

1. Unwilling or unable to discontinue use of contact lens during the study
2. Uncontrolled medical conditions that may in the judgment of the investigator confound the study assessments or limit compliance.
3. Known sensitivity to corticosteroids or a known "steroid responder"
4. Known hypersensitivity to the study drugs or the components or contraindications to hydrocortisone ophthalmic ointment
5. Use of any systemic or topical ophthalmic antihistamine agents within 72 hours before visit 1, and that cannot be discontinued during the study
6. Participation in an ophthalmic drug or device research study within 30 days prior to entry in this study.
7. Regular use of systemic or topical ophthalmic non-steroidal anti-inflammatory agents (NSAID), and analgesics
8. Younger than 18 years of age, Male or Female
9. Unwilling to provide written informed consent
10. Unlikely to complete all study visits
11. Patients diagnosed with Glaucoma
12. History of any ocular condition that, in the opinion of the investigator, could affect study parameters including, but not limited to, glaucoma, blepharitis, meibomian gland disease, follicular conjunctivitis, and/or active ocular infection or inflammation.
13. Use of any concurrent therapies for allergic conjunctivitis, prescription or over the counter.
14. Prohibited medications include:

    1. topical ophthalmic or systemic corticosteroids
    2. topical ophthalmic/nasal antihistamines (72 hour washout period prior to baseline/screening visit and no use throughout duration of the study)
    3. artificial tears/ocular lubricants (72 hour washout period and no use throughout the duration of the study)
    4. topical ophthalmic/nasal steroids (14 day washout period prior to baseline/screening visit and no use throughout the duration of the study) (Washout period can begin after Informed Consent Document is completed by the subject.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-05; Primary Completion 2016-05 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of Hydrocortisone Ophthalmic Ointment 0.5% vs. Placebo for the reduction of signs and symptoms associated with allergic conjunctivitis | 14 days
  Demonstration of efficacy is a statistically significant improvement in itching on a 0 to 4 patient subjective assessment itch score compared to the vehicle arm and at least a 25% (or 1 full unit or more) improvement in itch scores. Efficacy for bulbar redness scores would be indicated by a statistically significant improvement in redness on a zero to 4 based on the investigators objective assessment compared to the vehicle group. Differences of at least 25% on the four point scale would be considered clinically significant when attained at the majority of time points.

SECONDARY OUTCOMES:
Safety of Hydrocortisone Ophthalmic Ointment 0.5% vs. Placebo for the reduction of signs and symptoms associated with allergic conjunctivitis | 3 days, 14 days
  At each visit, the principal investigator or designated personnel determined to be medically qualified by the principal investigator will begin by querying for adverse events by asking each patient a general, non-directed question such as 'How have you been feeling since the last visit?' Directed questioning and examination will then be done as appropriate. All reported adverse events will be documented on the appropriate case report form.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Karpecki, OD, Principal Investigator — Clinical Research Director
Locations (1):
- Koffler Vision Group, Lexington, Kentucky, United States